CLINICAL TRIAL: NCT07243249
Title: Study Evaluating the Impact of Using Triplex Rapid Diagnostic Tests (SARS-CoV-2/Influenza/RSV) on Antibiotic Prescribing in the General Population in Community Settings
Brief Title: Study Evaluating the Impact of Using Triplex Rapid Diagnostic Tests (SARS-CoV-2/Influenza/RSV) on Antibiotic Prescribing
Acronym: TROD-VILLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: APHP250413; 2025-A02154-45 (Other: N° IDRCB)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Infections; Antibiotic
Keywords: Respiratory infections; Antibiotic; Rapid diagnostic tests
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients without triplex TROD tests. Doctors may or may not prescribe antibiotics probabilistically as usual.
- TROD (Experimental): Patient with triplex TROD test. Doctors may or may not prescribe antibiotics with the help of the results of triplex TROD tests.
  Interventions: Diagnostic Test: TROD

INTERVENTIONS:
Diagnostic Test: TROD — Patient with triplex TROD test. Doctors may or may not prescribe antibiotics with the help of the results of triplex TROD tests.
  Arms: TROD

SUMMARY:
Respiratory infections are very common, especially during winter, and are often caused by viruses such as influenza, SARS-CoV-2 or respiratory syncytial virus (RSV).

These illnesses are generally mild, but their symptoms do not always allow a clear distinction to be made between a viral infection and a bacterial infection. In the absence of a precise diagnosis, antibiotics may be prescribed when they are not necessary in many cases.

However, the excessive use of antibiotics contributes to the development of bacterial resistance, which is a major public health issue.

The aim of this study is to better understand whether the use of a rapid test (called TROD), which can quickly identify certain respiratory viruses, can help doctors reduce unnecessary antibiotic prescriptions for these infections. The test will be performed using a swab gently inserted into the nose.

DETAILED DESCRIPTION:
Bacterial resistance to antibiotics is a major global public health issue. In France, this resistance is estimated to cause 158,000 infections annually (127,000 to 245,000), including nearly 16,000 invasive infections, and 12,500 deaths per year. The additional cost of antibiotics in France compared to the average for the most virtuous European countries has been estimated at €441 million.

Reducing exposure to antibiotics by limiting their prescription to situations where they are essential is one of the major levers for slowing down the emergence of resistance.

The vast majority of antibiotics are prescribed in outpatient settings (90% of consumption, or 125 million units per year). In France, respiratory tract infections account for 7 out of 10 prescriptions in primary care. However, the majority of respiratory infections are viral in origin (influenza viruses, respiratory syncytial virus (RSV), SARS-CoV-2, but also rhinoviruses, metapneumoviruses, etc.). The clinical presentation of these infections is often non-specific. The lack of microbiological aetiological diagnosis leads to the unnecessary prescription of antibiotics in many cases of viral infections.

The rapid diagnostic tests (TROD) that have recently become available can test for RSV, influenza viruses and SARS-CoV-2 simultaneously. They enable a diagnosis of viral infection to be made during a consultation and should help to avoid the prescription of antibiotics in these situations. In addition, these tests are simple and can be performed routinely (in less than 15 minutes) without the need for specific equipment or technical skills. Reducing inappropriate prescriptions of antibiotic treatments for viral respiratory infections is therefore a public health priority that is likely to have a significant impact on bacterial resistance, but also on the incidence of adverse effects and the costs associated with these treatments.

At the request of the Haute Autorité de Santé (French National Authority for Health), this study aims to estimate the impact of triplex TRODs (SARS-CoV-2/ influenza/RSV detection) on antibiotic prescriptions in the general population in community settings among patients with infectious syndrome, and to produce data (comparative to RT-PCR) to better estimate the diagnostic performance, sensitivity and specificity of the test used in the study.

The participation period for each participating doctor will be determined by random draw, with the aim of ensuring that the start dates of participation are spread throughout the study period, and with each doctor having a first control period without the use of tests (n = 10 patients) followed by a second period with the use of tests (n = 10 patients). Antibiotic prescriptions will be collected for each patient included during the two periods.

Each investigator will begin the study (on the randomly selected date) by including 10 patients who meet the eligibility criteria during the period without testing (first period), then the investigating physician will move on to the second period and use the TROD for 10 other patients.

The main objective is to evaluate the impact of using triplex rapid diagnostic tests (SARS-CoV-2/influenza/RSV) on antibiotic prescribing in the general population in community settings during the autumn-winter season of 2025-2026.

The secondary objectives are to : 1. Compare the probability of prescription during the initial consultation between the two study periods, 2. Compare the frequency of patient re-consultations within 15 days of inclusion between the two study periods, 3. Compare the proportions of patients with secondary hospitalisation within 15 days of inclusion between the two study periods, 4. Compare total antibiotic consumption within 15 days of inclusion between the two study periods, 5. Conduct a cost-consequence medical-economic study, 6. Assess the impact of these tests according to patient characteristics (age, medical history, initial symptoms, etc.) and prescribers (age, geographical area, practice modalities.), 7. Assess the proportions of SARS-CoV-2/influenza/RSV during the intervention period in patients presenting with all of the described symptoms of respiratory infection, 8. Estimate the sensitivity and specificity of the TROD in identifying different viruses using respiratory multiplex PCR, as well as the frequency and nature of other respiratory viral infections, 9. Describe the epidemiology of other respiratory viral infections, whether or not associated with SARS-CoV-2/influenza/RSV infections.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 1 year
2. Presenting with:

   * Either fever (temperature > 38°C measured by patient or physician) within the past 72 hours, and one of the following symptom combinations:

     1. Rhinorrhea (white, yellow, or green discharge) and/or nasal obstruction, and cough
     2. Body aches, cough, and fatigue
     3. Odynophagia and negative strepto-test
     4. Cough
     5. Otalgia
   * Or suspicion of lower respiratory tract infection: signs of infection (respiratory rate > 20/min, heart rate > 100/min, fatigue, Body aches, chills, or fever), associated with pulmonary localization signs [cough, sputum, chest pain, auscultatory abnormality (rhonchi, crackles, or wheezing)]
3. Affiliation with the national health insurance system
4. Informed consent obtained from the adult participant, or from the person(s) with parental authority for a minor participant

Exclusion Criteria:

1. Requirement for hospitalization
2. Presence of a non-respiratory infection requiring concomitant antibiotic treatment.
3. Patients covered by State Medical Aid (AME)

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Variation in the probability of antibiotic prescription between adjacent periods differing in the use of tests TROD | Day 0 to Day 14
  Variation in antibiotic prescription rate between 1st periods during which doctors prescribe antibiotics probabilistically without rapid diagnostic tests (TROD) as usual, followed by 2nd periods during which antibiotic prescription is guided by the results of triple TROD (SARS-CoV-2/influenza/RSV). The primary endpoint will take into account all antibiotic prescriptions received by patients within 15 days of inclusion, whether they were prescribed at the end of the consultation that led to inclusion or during follow-up consultations.

SECONDARY OUTCOMES:
Percentage of patients receiving an antibiotic prescription at the initial consultation in both groups | Day 0
Percentage of patients requiring a new medical consultation between inclusion and day 14 in both groups | Day 0 to Day 14
Percentage of patients requiring secondary hospitalisation between inclusion and day 14 in both groups | Day 0 to Day 14
Total antibiotic consumption on day 14 in both groups | Day 0 to Day 14
Total cost of patient care | Day 0 to Day 14
  Cost-consequence medical-economic study
Previous criteria 2-4 according to patient characteristics and prescribers | Day 0 to Day 14
Percentage of patients with positive TROD results for the viruses studied during the intervention period (PCR and TROD) | Day 0 to Day 14
Estimation of the sensitivities and specificities of the TROD with regard to different viruses | Day 0
  TROD compared to the identification of different viruses using respiratory multiplex PCR in approximately 750 patients
Frequency of other respiratory viral infections associated or not associated with SARS-CoV-2/influenza/Respiratory syncytial virus infections | Day 0
  Epidemiology of other respiratory viral infections associated or not associated with SARS-CoV-2/influenza/RSV among Influenza A, Influenza B, Respiratory syncytial virus, SARS-CoV-2, Adenovirus B/E, Adenovirus C, Metapneumovirus, Enterovirus/rhinovirus, Coronavirus OC43, Coronavirus HKU1, Coronavirus 229E, Coronavirus NL63, Human parainfluenza virus 1 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien DINH, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Garches, France

IPD SHARING:
Plan to Share IPD: Undecided